CLINICAL TRIAL: NCT03098251
Title: Efficacy of 3D Typing and Routine Typing on Surgical Treatment of Hepatolithiasis
Brief Title: Effect of 3D Typing on Surgical Treatment of Hepatolithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, feng xiaobin, clinical professor, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWHB017
Record Dates: First submitted 2017-03-20; First posted 2017-03-31 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Hepatolithiasis; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D typing (Experimental): typing the patient with 3D typing system and give treatment according preestablished algorism in our center.
  Interventions: Procedure: 3D typing
- routine typing (Active Comparator): typing the patient with routine typing system and give treatment according preestablished algorism in our center.
  Interventions: Procedure: routine typing

INTERVENTIONS:
Procedure: 3D typing — typing the patient with 3D typing system and give specific treatment
  Arms: 3D typing
Procedure: routine typing — typing the patient with routine typing system and give specific treatment
  Arms: routine typing

SUMMARY:
According to a large amount of case affected with hepatolithiasis, we developed a typing system of Hepatolithiasis based on 3D digital conformation. And we hypothesized that it could predict a more precise construction of this disease, hence, typing by 3D conformation will improve the outcome of surgical treatment.The investigators will use a multicenter ambispective cohort study to test this hypothesis.

DETAILED DESCRIPTION:
According to a large amount of case affected with hepatolithiasis, we developed a typing system of Hepatolithiasis based on 3D digital conformation. And we hypothesized that it could predict a more precise construction of this disease, hence, typing by 3D conformation will improve the outcome of surgical treatment.The investigators will use a multicenter ambispective cohort study to test this hypothesis. In this cohort study, two group will be enrolled to compare the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 years old
* Without gender restriction
* With a favorable liver function of Child-Pugh A to B
* No contraindications to surgery and anesthesia
* Diagnosed with Hepatolithiasis and Signed informed consent.

Exclusion Criteria:

* Diffused type of Hepatolithiasis
* Impairment in liver function
* Severe disorders in vital organ
* Accompanied with tumors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
residual ratio of biliary stone | 3 months
  residual ratio of biliary stone diagnosed within 3 months

SECONDARY OUTCOMES:
postoperative complications | 6 months
  postoperative complications diagnosed within 6 months
residual lesions | 6 months
  residual lesions diagnosed within 6 months
Health economics index | 3 months
  Health economics index within 3 months
mortality | 3 months
  mortality occured within 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided